CLINICAL TRIAL: NCT04950764
Title: The Effect of Hepatic Impairment on The Pharmacokinetics of Seladelpar: An Open-Label Study Following Oral Dosing of Seladelpar to Subjects With Primary Biliary Cholangitis (PBC) and Hepatic Impairment
Brief Title: An Open-Label Study Following Oral Dosing of Seladelpar to Subjects With Primary Biliary Cholangitis (PBC) and Hepatic Impairment (HI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB8025-21838; 2020-005925-10 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2021-06-14; First posted 2021-07-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Primary Biliary Cholangitis; Compensated Cirrhosis; Hepatic Impairment
Keywords: PBC; Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — seladelpar

STUDY DESIGN:
Intervention Model Description: Seladelpar 10 mg
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seladelpar 10 mg (Experimental): Part A: Single oral dose 10 mg
  Interventions: Drug: Seladelpar 10 mg
- Seladelpar 10 mg or less (Experimental): Part B: Multiple oral dose of 10 mg or less
  Interventions: Drug: Seladelpar 10 mg or less

INTERVENTIONS:
Drug: Seladelpar 10 mg — Seladelpar 10 mg single oral dose
  Other Names: Livdelzi®
  Arms: Seladelpar 10 mg
Drug: Seladelpar 10 mg or less — Seladelpar 10 mg or less, once daily for 28 days
  Other Names: Livdelzi®
  Arms: Seladelpar 10 mg or less

SUMMARY:
The Effect of Hepatic Impairment on The Pharmacokinetics of Seladelpar: An Open-Label Study Following Oral Dosing of Seladelpar to Subjects with Primary Biliary Cholangitis (PBC) and Hepatic Impairment (HI)

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 80 years of age (inclusive) who are able to comprehend instructions and follow the study procedures and are willing to sign an Informed Consent Form (ICF)
2. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must be willing to use the contraceptive methods throughout the study and for 30 days after study drug administration.
3. For at least 90 days after study drug administration, non-vasectomized males must not donate sperm, be willing to use contraception with childbearing potential partners and any male subject with a pregnant partner must use a condom.
4. Willing to abstain from consuming grapefruit, pomelo, star fruit, or Seville orange containing products from 7 days prior to dose of study medication through day of discharge.
5. Confirmed diagnosis of PBC with evidence of cirrhosis and Child-Pugh classification of CP-A, CP-A + PHT, CP-B or CP-C
6. Screening laboratory parameters:

   * ALP, ALT and AST < 10 × ULN
   * Total bilirubin ≤ 5 × ULN
7. Ursodeoxycholic acid (UDCA) for a minimum of 12 weeks of treatment prior to Day 1
8. At screening confirmed diagnosis of PBC
9. MELD-Na scores of 6 to 24

Exclusion Criteria:

1. Clinically significant or history of acute or chronic liver disease of an etiology other than PBC
2. Patients with a diagnosis of overlapping PBC and autoimmune hepatitis
3. History, evidence, or high suspicion of hepatobiliary malignancy based on imaging, screening laboratory values, and/or clinical symptoms.
4. Presumptive or diagnosed infection that requires systemic therapy within 12 weeks of Screening and through Day 1
5. Female subjects who are pregnant or nursing
6. Screening ECG that demonstrates a QT interval ≥ 500 msec, or any other significant ECG finding with clinically significant abnormalities as determined by the Investigator
7. Positive for HBsAg, HCV RNA, or anti HIV antibody
8. Any non-hepatic acute or chronic condition that, in the opinion of the Investigator, would limit the patient's ability to complete and/or participate in the study or compromise the integrity of the data
9. Has experienced an illness that is considered by the Investigator to be clinically significant within 2 weeks before administration of investigational product
10. Clinically relevant drug or alcohol abuse within 6 months of Screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication
11. Use of obeticholic acid (OCA), any drug of the same class, or fibrates (e.g., bezafibrate, fenofibrate, elafibranor, lanifibranor, pemafibrate, saroglitizar) within 30 days of Baseline
12. Use of an experimental or unapproved treatment for PBC within 30 days of Baseline
13. Clinically evident complication(s) of cirrhosis and portal hypertension that required either emergency room visit, hospital admission or both during the 12 week period prior to investigational product administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluate maximum concentration (Cmax) of seladelpar and metabolites | 17 weeks
Evaluate the time to reach Cmax (Tmax) of seladelpar and metabolites | 17 weeks
Evaluate area under the concentration curve versus time curve of seladelpar and metabolites | 17 weeks
Evaluate the amount of seladelpar excreted in the urine (Ae) | 17 weeks
Evaluate safety and tolerability as assessed by the incidence of treatment emergent adverse events and serious treatment emergent adverse events across child pugh treatment groups | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (20):
- United States (11):
  - Arizona Liver Health, Chandler, Arizona
  - University of California Davis, Sacramento, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Weill Medical College of Cornell University, New York, New York
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research- SA, San Antonio, Texas
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Hospital General Universitario Gregorio Maran, Madrid, Spain
- United Kingdom (3):
  - NIHR BRC Centre for Liver and Gastrointestinal Research Birmingham, Birmingham
  - The Royal Free London NHS Foundation Trust, London
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No